CLINICAL TRIAL: NCT06008197
Title: Randomized Trial to Determine the Efficacy and Safety of Finerenone on Morbidity and Mortality Among Heart Failure Patients With Left Ventricular Ejection Fraction Greater Than or Equal to 40% Hospitalized Due to an Episode of Acute Decompensated Heart Failure (REDEFINE-HF)
Brief Title: A Study to Determine the Efficacy and Safety of Finerenone on Morbidity and Mortality Among Hospitalized Heart Failure Patients
Acronym: REDEFINE-HF
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Colorado Prevention Center (Other)
Collaborators: St. Luke's Hospital, Kansas City, Missouri (Other); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202301CPC
Record Dates: First submitted 2023-07-31; First posted 2023-08-23 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure; Acute Heart Failure
Keywords: Heart failure; Preserved ejection fraction; Mildly reduced ejection fraction; Hospitalized
MeSH Terms: conditions — Heart Failure | interventions — finerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Finerenone (Experimental)
  Interventions: Drug: Finerenone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Finerenone — Oral finerenone
  Other Names: Kerendia
  Arms: Finerenone
Drug: Placebo — Matching oral placebo
  Arms: Placebo

SUMMARY:
Finerenone will be compared to placebo to determine efficacy and safety of treatment in patients hospitalized with acute decompensated heart failure (HF) and mildly reduced or preserved left ventricular ejection fraction.

DETAILED DESCRIPTION:
This is an international, randomized, double-blind, placebo-controlled, event-driven trial of finerenone for the treatment hospitalized heart failure patients with mildly reduced or preserved ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

* Provide electronic or written informed consent, either personally or through a legally authorized representative
* Age ≥18 years
* Current hospitalization or recently discharged with the primary diagnosis of heart failure
* Heart failure signs and symptoms at the time of hospital admission
* Imaging evidence of mildly reduced or preserved left ventricular ejection fraction (EF) (40% or higher)
* Elevated N-terminal pro B-type natriuretic peptide (NTproBNP) ≥1000 pg/mL or B-type natriuretic peptide (BNP) ≥250 pg/mL for patients without atrial fibrillation (AF); or elevated NTproBNP ≥2000 pg/mL or BNP ≥500 pg/mL for patients with AF

Exclusion Criteria:

* Treatment with a mineralocorticoid receptor antagonist (MRA)
* Documented prior history of severe hyperkalemia in the setting of MRA use
* Estimated glomerular filtration rate (eGFR) <25 mL/min/1.73m² or serum/plasma potassium >5.0 mmol/L at screening
* Acute myocardial infarction, coronary revascularization, valve replacement/repair, or implantation of a cardiac resynchronization therapy device within 30 days
* Hemodynamically significant (severe) uncorrected primary cardiac valvular disease
* Cardiomyopathy due to known acute inflammatory heart, infiltrative diseases, accumulation diseases, muscular dystrophies, cardiomyopathy with reversible causes, known hypertrophic obstructive cardiomyopathy, complex congenital heart disease, or known pericardial constriction
* Probable alternative cause of participant's heart failure symptoms
* Concomitant systemic therapy with potent cytochrome P450 isoenzyme 3A4 (CYP3A4) inhibitors or moderate CYP3A4 inducers, or potent CYP3A4 inducers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5200 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Composite total of HF events and cardiovascular (CV) death. | Ongoing, up to ~30 months
  Total (first and subsequent) HF hospitalizations, urgent visits for worsening HF, and CV deaths with finerenone compared to placebo.
Number of serious adverse events. | Ongoing, up to ~30 months
  Occurrence of serious adverse events (excluding efficacy endpoints) with finerenone compared to placebo.
Number of adverse events leading to discontinuation of study drug. | Ongoing, up to ~30 months
  Occurrence of adverse events leading to study drug discontinuation with finerenone compared to placebo.

SECONDARY OUTCOMES:
Time to first occurrence of the composite of CV death or HF event. | Ongoing, up to ~30 months
  Time to first occurrence of the composite of CV death or HF event with finerenone compared to placebo.
Total HF events. | Ongoing, up to ~30 months
  Total HF events with finerenone compared to placebo.
Change from baseline in the Total Symptom Score on the Kansas City Cardiomyopathy Questionnaire (KCCQ-TSS) at Month 6. | 6 Months
Time to CV death. | Ongoing, up to ~30 months
  Time to CV death with finerenone compared to placebo.
Time to death from any cause. | Ongoing, up to ~30 months
  Time to death from any cause with finerenone compared to placebo.

OTHER OUTCOMES:
Total hospitalizations for any cause. | Ongoing, up to ~30 months
  Total hospitalizations for any cause with finerenone compared to placebo.
Total number of days alive and out of the hospital. | Ongoing, up to ~30 months
  Days alive and out of hospital with finerenone compared to placebo.
Number of patients with sustained decrease in eGFR ≥40% relative to baseline. | Ongoing, up to ~30 months
  Sustained decrease in eGFR ≥40% relative to baseline with finerenone compared to placebo.
Number of patients with sustained eGFR <15 ml/min/1.73 m^2. | Ongoing, up to ~30 months
  Sustained eGFR <15 ml/min/1.73 m^2 with finerenone compared to placebo.
Number of patients requiring initiation of dialysis or renal transplant. | Ongoing, up to ~30 months
  Initiation of dialysis or renal transplant with finerenone compared to placebo.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Aurora, CO Investigative Site, Aurora, Colorado
  - Denver, CO Investigative Site, Denver, Colorado
  - Boca Raton, FL Investigative Site, Boca Raton, Florida
  - Kansas City, MO Investigative Site, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No
No current plan to share individual patient data with other researchers.